CLINICAL TRIAL: NCT04000815
Title: Serum Levels of C Type Natriuretic Peptide in Reproductive Age, Perimenopausal and Postmenopausal Women
Brief Title: Serum Levels of C Type Natriuretic Peptide in Different Reproductive Periods
Acronym: CO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Ali Cenk, Medical Doctor, Near East University, Turkey
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CenkOzay
Record Dates: First submitted 2019-06-22; First posted 2019-06-27 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Serum CNP Levels; Healthy Reproductive Age Women; Healthy Perimenopausal Women; Healthy Postmenopausal Women
Keywords: c type natriuretic peptide; duration of menopause; menstrual cycle

STUDY DESIGN:
Intervention Model Description: In this study, there are three groups. Group 1:Women between 18-40 age, Group 2:Perimenopausal women (40-49 years), Group 3: Postmenopausal women.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reproductive age women (Active Comparator): The healthy women between 18-40 years old.
  Interventions: Diagnostic Test: C Type Natriüretic Peptide
- Perimenopausal women (Active Comparator): The healthy women between 40-49 years old.
  Interventions: Diagnostic Test: C Type Natriüretic Peptide
- Postmenopausal women (Active Comparator): The healthy women that has been in to menopause more than a year
  Interventions: Diagnostic Test: C Type Natriüretic Peptide

INTERVENTIONS:
Diagnostic Test: C Type Natriüretic Peptide — C Type Natriuretic Peptide will be measured with elisa method

SUMMARY:
Recent studies have shown that C natriuretic peptide (CNP) is produced from granulosa cells, increasing cumulative guanosine monophosphate (cGMP) production by affecting cumulus cells through natriuretic peptide receptors.It has been suggested that the transport of cGMP to oocyte via gap junctions causes a continuous increase in cyclic adenosine monophosphate (cAMP) levels within the oocyte. An important role of increased cAMP levels in oocyte is shown to suppress meiotic progression. Deoxyribonucleic acid (DNA) studies in animals have shown that expression of the natriuretic peptide precursor increases during the periovulatory period and shows that this increase decreases rapidly after Luteinizing hormone(LH) / human chorionic(hCG) stimulation. Human studies have shown that after ovulation induction, the CNP level in follicular fluid decreases following ovulatory dose of hCG (9).

DETAILED DESCRIPTION:
In this prospective study, 60 patients are planned to recruite. Group 1 consists of 20 healthy reproductive aged women between 18-40 years old, with regular menstruation. Group 2 will include 20 patients in perimenopausal time period between 40-49 ages and in group 3 there will be20 postmenopausal women.

Age, gravida, parity and body mass index (BMI) data of all patients will be recorded. BMI is calculated by dividing the body weight in kilograms by the square of the height in meters. All patients will go under ultrasound examination by the same clinician (ACO). The number of antral follicles in group 1 and group 2 will be recorded. In addition, on the 2nd or 3rd day of menstruation, serum FSH, LH and E2 data of the patients in group 1 and 2 will be recorded.

For the last 6 months, patients with drug use that may affect menstruation like oral contraceptives, patients with cardiac or renal disease and therefore drug use, causes of infertility other than unexplained infertility, history of ovarian surgery, presence of polycystic ovary syndrome, and patients with irregular menstruation will be excluded for the study. In addition, patients with renal, cardiac, central nervous system and endocrine diseases will be excluded.

Morning fasting venous blood samples will be taken from the patients on the 2nd or 3rd day of the menstruation for group 1 and 2. All blood samples will be centrifuged on the day of collection and separated serum samples and will be kept at -80 degrees until the day of CNP test. Serum CNP levels of the patients will be analyzed by an enzyme-linked immunosorbent (ELISA) assay for human CNP in accordance with the manufacturer's instructions (SEA721Hu, ELISA Kit for Human CNP, Wuhan USCN Business Co., Ltd., Cloud-Clone Corp., CCC, USA).

Data will be analyzed using Statistical Package for Social Sciences software (SPSS v15, SPSS Inc, Chicago, IL, USA). The variables will be investigated using visual and analytical methods (histograms, homogeneity of variances test, Kolmogorov-Simirnov/Shapiro-Wilk's test) to determine whether or not they are normally distributed. Patient demographics and CNP values will be presented as median ± interquartile range. Gravida and parity will be demonstrated by frequency distribution. The correlation coefficients and their significance will be calculated using the Spearman test. P-values less than 0.05 will be regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Regular cyclic menstruation for reproductive age group

Exclusion Criteria:

* No systemic disease(cardiac, renal...etc)
* Smoking
* Drug usage
* Pregnancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants will be included
Enrollment: 71 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Özay, Principal Investigator — Near East University
Locations (1):
- Near East University Faculty of Medicine, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
Only the name of study

REFERENCES:
- [Background] Zhang M, Su YQ, Sugiura K, Xia G, Eppig JJ. Granulosa cell ligand NPPC and its receptor NPR2 maintain meiotic arrest in mouse oocytes. Science. 2010 Oct 15;330(6002):366-9. doi: 10.1126/science.1193573. PMID 20947764
- [Background] Norris RP, Ratzan WJ, Freudzon M, Mehlmann LM, Krall J, Movsesian MA, Wang H, Ke H, Nikolaev VO, Jaffe LA. Cyclic GMP from the surrounding somatic cells regulates cyclic AMP and meiosis in the mouse oocyte. Development. 2009 Jun;136(11):1869-78. doi: 10.1242/dev.035238. PMID 19429786
- [Background] Vaccari S, Weeks JL 2nd, Hsieh M, Menniti FS, Conti M. Cyclic GMP signaling is involved in the luteinizing hormone-dependent meiotic maturation of mouse oocytes. Biol Reprod. 2009 Sep;81(3):595-604. doi: 10.1095/biolreprod.109.077768. Epub 2009 May 27. PMID 19474061
- [Background] Tsafriri A, Chun SY, Zhang R, Hsueh AJ, Conti M. Oocyte maturation involves compartmentalization and opposing changes of cAMP levels in follicular somatic and germ cells: studies using selective phosphodiesterase inhibitors. Dev Biol. 1996 Sep 15;178(2):393-402. doi: 10.1006/dbio.1996.0226. PMID 8812137
- [Background] Thomas RE, Armstrong DT, Gilchrist RB. Differential effects of specific phosphodiesterase isoenzyme inhibitors on bovine oocyte meiotic maturation. Dev Biol. 2002 Apr 15;244(2):215-25. doi: 10.1006/dbio.2002.0609. PMID 11944932
- [Background] Nogueira D, Albano C, Adriaenssens T, Cortvrindt R, Bourgain C, Devroey P, Smitz J. Human oocytes reversibly arrested in prophase I by phosphodiesterase type 3 inhibitor in vitro. Biol Reprod. 2003 Sep;69(3):1042-52. doi: 10.1095/biolreprod.103.015982. Epub 2003 May 28. PMID 12773402
- [Background] Lee KB, Zhang M, Sugiura K, Wigglesworth K, Uliasz T, Jaffe LA, Eppig JJ. Hormonal coordination of natriuretic peptide type C and natriuretic peptide receptor 3 expression in mouse granulosa cells. Biol Reprod. 2013 Feb 21;88(2):42. doi: 10.1095/biolreprod.112.104810. Print 2013 Feb. PMID 23255339
- [Background] Hiradate Y, Hoshino Y, Tanemura K, Sato E. C-type natriuretic peptide inhibits porcine oocyte meiotic resumption. Zygote. 2014 Aug;22(3):372-7. doi: 10.1017/S0967199412000615. Epub 2013 Jan 18. PMID 23331536
- [Background] Kawamura K, Cheng Y, Kawamura N, Takae S, Okada A, Kawagoe Y, Mulders S, Terada Y, Hsueh AJ. Pre-ovulatory LH/hCG surge decreases C-type natriuretic peptide secretion by ovarian granulosa cells to promote meiotic resumption of pre-ovulatory oocytes. Hum Reprod. 2011 Nov;26(11):3094-101. doi: 10.1093/humrep/der282. Epub 2011 Aug 23. PMID 21865234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the last 6 months, patients with drug use that may affect menstruation like oral contraceptives, patients with cardiac or renal disease and therefore drug use, causes of infertility other than unexplained infertility, history of ovarian surgery, presence of polycystic ovary syndrome, and patients with irregular menstruation.
Period: Overall Study
Arm/Group | Reproductive Age Women | Perimenopausal Women | Postmenopausal Women
Started | 29 | 20 | 22
Completed | 15 | 15 | 15
Not Completed | 14 | 5 | 7
Not completed — Lost to Follow-up | 9 | 2 | 3
Not completed — Withdrawal by Subject | 4 | 3 | 2
Not completed — Right ovarian cyst occured | 1 | 0 | 0
Not completed — Hypertension occured on follow up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproductive Age Women | Perimenopausal Women | Postmenopausal Women | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (2.9) | 44.1 (2.2) | 57.7 (5.4) | 42.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 45
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Cyprus | 15 | 15 | 15 | 45
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.3 (1.9) | 24.3 (2.4) | 27.1 (4.1) | 24.2 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Serum C Type Natriuretic Peptide Levels
Description: The comparison of serum levels of C type natriuretic peptide among different age groups
Time Frame: Second or Third Day of Menstruation
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Reproductive Age Women | Perimenopausal Women | Postmenopausal Women
Number analyzed (Participants) | 15 | 15 | 15
pg/ml | 43.68 [35.54 to 47.87] | 55.98 [49.84 to 61.14] | 116.36 [59.61 to 250.00]
Statistical Analysis 1: Comparison: Reproductive Age Women vs Perimenopausal Women vs Postmenopausal Women; Test type: Other; p < 0.017, Kruskal-Wallis — p-value is adjusted for multiple comparisons

2. Secondary Outcome: Correlation Between Serum CNP and Follicle Stimulating Hormone and Luteinizing Hormone Levels in Groups 1 and 2
Description: Correlations between serum CNP vs Follicle Stimulating Hormone(FSH), CNP vs Luteinizing Hormone(LH) levels in groups 1 and 2
Time Frame: Second or Third Day of Menstruation
Population: FSH and LH should be evaluated during menstruation time period ( day 3). In postmenopausal women there is no spesific date to evaluate these hormones since they do not have menstruation. Therefore in postmenopausal arm group these hormones (FSH and LH) are not studied.
Measure: Median (Inter-Quartile Range); unit: mIU/mL
Arm/Group | Reproductive Age Women | Perimenopausal Women
Number analyzed (Participants) | 15 | 15
mIU/mL
  Follicle Stimulating Hormone | 5.28 [4.68 to 6.01] | 13.12 [9.15 to 16.45]
  Luteinizing Hormone | 5.71 [4.62 to 7.13] | 5.16 [3.75 to 6.20]
Statistical Analysis 1: Comparison: Reproductive Age Women vs Perimenopausal Women; Test type: Other; p < 0.05, Bi-variate correlation analysis; Bi-variate correlation analyses were performed in groups 1 and 2 between serum CNP and FSH and between serum CNP and LH using Spearman test

3. Secondary Outcome: Correlation Between Serum CNP and Antral Follicle Count (AFC) in Groups 1 and 2
Description: Correlation between serum CNP and antral follicle count (AFC) in groups 1 and 2 using Spearman test
Time Frame: Second or Third Day of Menstruation
Population: AFC should be evaluated during menstruation time period ( day 3). In postmenopausal women there is no spesific date to evaluate AFC value since they do not have menstruation. Therefore in postmenopausal arm group AFC value is not studied.
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Reproductive Age Women | Perimenopausal Women
Number analyzed (Participants) | 15 | 15
follicles | 14.2 (2.18) | 8.33 (1.72)
Statistical Analysis 1: Comparison: Reproductive Age Women vs Perimenopausal Women; Test type: Other; p < 0.05, Bi-variate correlation; Spearman test was applied

4. Secondary Outcome: Correlation Between Serum CNP and Estradiol Levels in Groups 1 and 2
Description: Correlation of CNP vs. Estradiol levels in reproductive age and perimenopausal women
Time Frame: Second or Third Day of Menstruation
Population: Estradiol should be evaluated during menstruation time period ( day 3). In postmenopausal women there is no spesific date to evaluate this hormone since they do not have menstruation. Therefore in postmenopausal arm group this hormone is not studied.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Reproductive Age Women | Perimenopausal Women
Number analyzed (Participants) | 15 | 15
pg/mL | 41 [33 to 59] | 22 [16 to 30]
Statistical Analysis 1: Comparison: Reproductive Age Women vs Perimenopausal Women; Test type: Other; p < 0.05, Bi-variate correlation analyses; Bi-variate correlation analyses were performed for all subjects in groups 1 and 2 between serum CNP and E2 using Spearman test

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed.
Description: Adverse events were not assessed.
Arm/Group | Reproductive Age Women | Perimenopausal Women | Postmenopausal Women
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The most prominent limitation of our study was the relatively small number of participants. This avoided us from using more powerful parametric tests for statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT04000815/Prot_SAP_000.pdf